CLINICAL TRIAL: NCT02254772
Title: A Phase I/II Study of Intratumoral Injection of SD-101, an Immunostimulatory CpG, and Intratumoral Injection of Ipilimumab, an Anti-CTLA4 Monoclonal Antibody, in Combination With Local Radiation in Low-Grade B-Cell Lymphomas
Brief Title: A Phase I/II Study of Intratumoral Injection of SD-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Robert Lowsky (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Lowsky, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-31133; NCI-2014-01978 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LYMNHL0119 (Other: OnCore number); 5R01CA188005-02 (NIH)
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2017-02

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Ipilimumab; CTLA-4 Antigen; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients receive TLR9 agonist SD-101 via intratumoral injections; ipilimumab via intratumoral injection; and undergo radiation therapy on days 1 and 2.
  Interventions: Biological: Ipilimumab; Drug: SD-101; Radiation: Radiation therapy

INTERVENTIONS:
Biological: Ipilimumab — A dose of 10 mg in cohort 1 or 25mg in cohort 2 via intratumoral injection on day 2, week 1.
  Other Names: Yervoy; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4
Drug: SD-101 — Started on day 2 week 1, then once every week x 4 successive weeks for a total of 5 injections.
  Other Names: ISS-ODN SD-101; TLR9 agonist
Radiation: Radiation therapy — Undergo low-dose radiation therapy to 1 site of disease
  Other Names: Irradiation; Radiotherapy

SUMMARY:
This phase 1-2 trial studies the side effects and best dose of ipilimumab in combination with toll-like receptor 9 (TLR9) agonist SD-101 and radiation therapy in treating patients with recurrent low-grade B-cell lymphoma.

DETAILED DESCRIPTION:
Monoclonal antibodies, such as ipilimumab, may block cancer growth in different ways by targeting certain cells. Biological therapies, such as TLR9 agonist SD-101, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Giving ipilimumab in combination with TLR9 agonist SD-101 and radiation therapy may be a better treatment for B-cell lymphoma.

Study objectives are dose-limiting toxicity (DLT) and the treatment assessments tumor response and time-to-progression. Cohort 1 dose level is 10 mg ipilimumab, subsequent cohort is 5 or 25 mg ipilimumab.

* If 2 out of 6 patients experience a DLT in the first cohort (10 mg ipilimumab), the dose will be de-escalated to 5 mg ("Cohort -1").
* If 2 out of 6 patients experience a DLT at the 5 mg dose level, then the study will be stopped.

ELIGIBILITY:
Inclusion Criteria

* Biopsy-confirmed low-grade B-cell lymphoma, specifically, follicular grade 1 or 2, or 3A marginal zone or small lymphocytic lymphoma; patients must have relapsed from or are refractory to prior therapy
* Patients must have at least one site of disease that is accessible for intratumoral injection of SD-101 and of ipilimumab (diameter ≥ 10mm), percutaneously
* Tumor specimens must be available for immunological studies either from a previous biopsy or a new biopsy obtained before the initiation of the study
* Patients must have measurable disease other than the injection site or biopsy site
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 [corresponds to Karnofsky Performance Status (KPS) of ≥ 70]
* White blood cell count (WBC) ≥ 2000/µL (2 x 10^9/L)
* Absolute neutrophil count (ANC) ≥ 1000/µL (0.5 x 10^9/L)
* Platelets ≥ 75 x 10^3/µL (75 x 10^9/L)
* Hemoglobin ≥ 8 g/dL (may be transfused)
* Creatinine ≤ 2.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 x ULN for subjects without liver metastasis; ≤ 5 times for liver metastases
* Bilirubin ≤ 2.0 x ULN (except for subjects with Gilbert's Syndrome, who must have a total bilirubin of less than 3.0 mg/dL)
* No active or chronic infection with human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C
* Must be at least 4 weeks since treatment with standard or investigational chemotherapy, biochemotherapy, surgery, radiation, cytokine therapy, and 8 weeks since any monoclonal antibodies or immunotherapy, and recovered from any clinically significant toxicity experienced during treatment
* Patients of reproductive potential must agree to use an effective (> 90% reliability) form of contraception during the study and for 6 months following the last study drug administration
* Women of reproductive potential must have negative urine pregnancy test
* Life expectancy greater than 4 months
* Able to comply with the treatment schedule
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

* Pre-existing autoimmune or antibody mediated disease including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, Addison's disease, but excluding the presence of auto-antibodies without clinical autoimmune disease
* History of inflammatory bowel disease (eg, Crohn's disease or ulcerative colitis), celiac disease, or other chronic gastrointestinal conditions associated with diarrhea, or current acute colitis of any origin
* Any history of diverticulitis, or evidence of diverticulitis at baseline, including evidence limited to computed tomography (CT) scan only (note diverticulosis is not an exclusion criterion)
* Severe psoriasis
* Active thyroiditis
* History of uveitis
* Known history of HIV; patients with Acquired Immunodeficiency Syndrome (AIDS) are excluded
* Patients with active infection or with a fever > 38.5 degrees C within 3 days prior to the first scheduled treatment
* Central nervous system (CNS) lymphoma
* Prior malignancy (active within 5 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix
* History of allergic reactions attributed to compounds of similar composition to SD-101 or ipilimumab (anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA4] antibodies)
* Current anticoagulant therapy (EXCEPTION acetylsalicylic acid ≤ 325 mg per day allowed)
* Treatment with an immunosuppressive regimen of corticosteroids or other immunosuppressive medication (eg, methotrexate, rapamycin) within 30 days of study treatment; note patients with adrenal insufficiency may take up to 5 mg of prednisone or equivalent daily; topical and inhaled corticosteroids in standard doses are allowed
* Significant cardiovascular disease [ie, New York Heart Association (NYHA) class 3 congestive heart failure; myocardial infarction with the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias]
* Pregnant or lactating
* Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-09; Primary Completion 2016-11-10 (Actual); Study Completion 2017-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, MD, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185
- [Derived] Mooney KL, Czerwinski DK, Shree T, Frank MJ, Haebe S, Martin BA, Testa S, Levy R, Long SR. Serial FNA allows direct sampling of malignant and infiltrating immune cells in patients with B-cell lymphoma receiving immunotherapy. Cancer Cytopathol. 2022 Mar;130(3):231-237. doi: 10.1002/cncy.22531. Epub 2021 Nov 15. PMID 34780125

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (SD-101 + Ipilimumab + Radiation): Patients receive TLR9 agonist SD-101 via intratumoral injections; ipilimumab via intratumoral injection; and undergo radiation therapy on days 1 and 2.
Period: Overall Study
Arm/Group | Treatment (SD-101 + Ipilimumab + Radiation)
Started | 9
Completed | 7
Not Completed | 2
Not completed — Ineligible | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (SD-101 + Ipilimumab + Radiation)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose-limiting Toxicity (DLT) Events of Ipilimumab Plus a Fixed Dose of SD-101 (1 mg/Week)
Description: To determine the safety and tolerability of SD-101 (1 mg/week) and local low dose radiation plus escalating doses of subcutaneously (SC)-administered ipilimumab, the incidence of dose-limiting toxicities (DLT) will be assessed according to the following DLT definitions. Related adverse events (AEs) are toxicities. "Treatment" includes radiation therapy.
  * Grade 4 treatment-related AE
  * Any drug-related AE ≥ Grade 3, including injection site reaction
  * ≥ Grade 3 treatment-related clinical autoimmune reaction involving major organs (defined as liver, pancreas, lung, heart, kidney, bowel, bone marrow, eye, or central nervous system) which does not resolve to baseline or Grade 1 within 6 weeks
  * Treatment-related AE ≥ Grade 3 that persists despite adequate/maximal medical therapy and/or prophylaxis, EXCEPT
    * Treatment-related skin rash ≤ Grade 3, that does not require systemic steroid therapy or other immunosuppressive therapy OR
    * Grade 3 flu-like AEs
  * Uveitis ≥ Grade 2
Time Frame: Up to 10 weeks
Population: Only the starting dose level of 10 mg ipilimumab plus SD-101 (1 mg/week) was evaluated. The dose level of ipilimumab could not be escalated due to inability to obtain a higher concentration of ipilimumab.
Measure: Number; unit: Dose-limiting toxicity events
Arm/Group | Treatment (SD-101 + Ipilimumab + Radiation)
Number analyzed (Participants) | 7
Dose-limiting toxicity events | 0

2. Secondary Outcome: Tumor Response
Description: Tumor response was assessed per the Cheson Criteria for low-grade B-cell lymphomas.
  Complete Response (CR) - No evidence disease. Partial Response (PR) - Regression of measurable disease with no new sites Progressive Disease (PD) - Any new lesion or increase by ≥ 50% of any previously-involved site after treatment nadir.
  Stable Disease (SD) - Any status that is not CR; PR; or PD. See references (Cheson BD, et al. J Clin Oncol. Apr 1999;17(4):1244. PubMed ID 10561185.
Time Frame: Up to 2 years
Population: Note that 1 participants initially experienced a partial response (PR), but later had progressive disease (PD).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SD-101 + Ipilimumab + Radiation)
Number analyzed (Participants) | 7
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 6

3. Secondary Outcome: Median Time to Progression (TTP)
Description: Tumor progression was assessed as any new lesion or increase by ≥ 50% of any previously-involved site after treatment nadir.
Time Frame: Up to 2 years
Population: 1 participant had stable disease, but did not provide a final follow-up at 2 years.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (SD-101 + Ipilimumab + Radiation)
Number analyzed (Participants) | 6
Months | 3.33 [0.53 to 12.32]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (SD-101 + Ipilimumab + Radiation)
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SD-101 + Ipilimumab + Radiation) (N=9)
Neutropenia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SD-101 + Ipilimumab + Radiation) (N=9)
Neutropenia (Infections and infestations) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 9 (13)
Fever (General disorders) | 5 (5)
Injection site reaction (General disorders) | 5 (5)
Swelling (General disorders) | 3 (3)
Chills (General disorders) | 4 (4)
Flu Like Symptoms (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Increased Creatinine (Investigations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (11)
Induration (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Reproductive system and breast disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No